CLINICAL TRIAL: NCT00814359
Title: A Phase III Study of Magic Mouthwash Plus Sucralfate Versus Benzydamine HCl for Treatment of Radiation-induced Oral Mucositis in Head and Neck Cancer Patients.
Brief Title: Magic Mouthwash Plus Sucralfate Versus Benzydamine Hydrochloride for the Treatment of Radiation-induced Mucositis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Dr. Joda Kuk, Principal Investigator, Juravinski Cancer Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUCOSA-PROTECT
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2009-05

CONDITIONS: Head and Neck Cancer; Mucositis
Keywords: mucositis; radiation; magic mouthwash; sucralfate; benzydamine; diphenhydramine; dexamethasone; nystatin
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis | interventions — Sucralfate; Benzydamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magic Mouthwash Plus Sucralfate (Experimental)
  Interventions: Drug: Combination of Magic Mouthwash Plus Sucralfate
- Benzydamine HCl (Active Comparator)
  Interventions: Drug: 0.15% Benzydamine HCl

INTERVENTIONS:
Drug: Combination of Magic Mouthwash Plus Sucralfate — Magic mouthwash will contain diphenhydramine powder 375mg, dexamethasone injection 2.8mg, and nystatin suspension 50ml (1000 units/ml) diluted to a total volume of 250ml with sterile water.
  The concentration of the sucralfate suspension will be 1g/5ml.
  Patients will be instructed to rinse first with 5ml of the magic mouthwash solution for 2 minutes then swallow, followed by rinsing with 5ml of the sucralfate suspension for 2 minutes before swallowing, repeating this 4 times daily, starting on the day prior to the initiation of radiotherapy, and stopping 2 weeks after the completion of radiotherapy.
  Other Names: Mucositis Mouthwash; Sulcrate
  Arms: Magic Mouthwash Plus Sucralfate
Drug: 0.15% Benzydamine HCl — Patients will rinse with 15ml of 1.5mg/ml benzydamine HCl for 2 minutes then expectorate the solution, repeating this 4 times daily, starting on the day prior to the initiation of radiotherapy, and stopping 2 weeks after the completion of radiotherapy.
  Other Names: Tantum
  Arms: Benzydamine HCl

SUMMARY:
Radiation treatment is very effective for treating cancers of the head and neck, however, during the course of treatment, it is common for patients to experience soreness of their mouth and throat due to the radiation. When radiation causes inflammation of the inside of the mouth, it is called 'mucositis'. There are several mouthwashes that are commonly used to prevent and treat mucositis, but none of these have been shown to be superior to another. This study is being conducted to see if using a combination of magic mouthwash and sucralfate is better than using a single mouthwash called benzydamine at decreasing the burden of mucositis.

DETAILED DESCRIPTION:
Sixty patients with head and neck cancer being treated with 6 or more weeks of radiotherapy, will be randomly assigned to receive either a combination of magic mouthwash (diphenhydramine, dexamethasone and nystatin) plus sucralfate or benzydamine. Patients randomized to receive magic mouthwash plus sucralfate will rinse first with 5ml of the magic mouthwash for 2 minutes then swallow, followed by rinsing with 5ml of the 1g/5ml sucralfate for 2 minutes before swallowing, 4 times daily. Patients randomized to receive 0.15% benzydamine HCl will be instructed to rinse with 15ml of the solution for 2 minutes before expectorating, 4 times daily. Patients will start the mouthwash regimens prior to the initiation of radiotherapy, and stop 2 weeks after the completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the head and neck.
* Receiving 6 or more weeks of external beam radiotherapy to a treatment volume that includes mucosal surfaces of the head and neck.

Exclusion Criteria:

* Age less than 18 years
* ECOG Performance Score 2 or higher
* Patient is unable to understand the protocol and/or unable to provide informed consent
* Patient is unable or unwilling to complete the questionnaires which are written in English.
* Prior radiation to the head and neck region that would result in overlap of fields for the current study.
* Plan to receive a radiation treatment volume that only includes the larynx and or hypopharynx with no planned treatment of locoregional lymph nodes.
* Plan to receive a concurrent chemotherapy agent other than cisplatin.
* Plan to receive other investigational agents (eg. panitumumab).
* Investigational agent of any kind within 30 days prior to randomization.
* Concurrent administration of any other experimental intervention given for the purpose of preventing oral mucositis.
* History of allergic or hypersensitivity reactions to any of the possible agents to be administered in the study.
* Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The severity of patient-reported symptoms of mucositis as determined by the change in Oral Mucositis Weekly Questionnaire - Head and Neck Cancer (OMWQ-HN) score from baseline to 6 weeks. | Baseline to 6 weeks after the initiation of radiotherapy.

SECONDARY OUTCOMES:
The severity of patient-reported symptoms of mucositis throughout the course radiotherapy as determined by the area under the curve for mean change in OMWQ-HN scores from baseline. | Baseline to 10 weeks after initiating radiotherapy.
Incidence of WHO Grade 3 or 4 oral mucositis after 4 weeks of radiotherapy. | 4 weeks after initiating radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Joda Kuk, MD, Principal Investigator — Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Epstein JB, Silverman S Jr, Paggiarino DA, Crockett S, Schubert MM, Senzer NN, Lockhart PB, Gallagher MJ, Peterson DE, Leveque FG. Benzydamine HCl for prophylaxis of radiation-induced oral mucositis: results from a multicenter, randomized, double-blind, placebo-controlled clinical trial. Cancer. 2001 Aug 15;92(4):875-85. doi: 10.1002/1097-0142(20010815)92:43.0.co;2-1. PMID 11550161
- [Background] Epstein JB, Beaumont JL, Gwede CK, Murphy B, Garden AS, Meredith R, Le QT, Brizel D, Isitt J, Cella D. Longitudinal evaluation of the oral mucositis weekly questionnaire-head and neck cancer, a patient-reported outcomes questionnaire. Cancer. 2007 May 1;109(9):1914-22. doi: 10.1002/cncr.22620. PMID 17377917
- [Background] Wright JR, McKenzie M, DeAngelis C, Foroudi F, Paul N, Rajaraman M, Wong F, Wong R, Wong KS. Radiation induced mucositis: co-ordinating a research agenda. Clin Oncol (R Coll Radiol). 2003 Dec;15(8):473-7. doi: 10.1016/j.clon.2003.07.002. PMID 14690003
- [Background] Sutherland SE, Browman GP. Prophylaxis of oral mucositis in irradiated head-and-neck cancer patients: a proposed classification scheme of interventions and meta-analysis of randomized controlled trials. Int J Radiat Oncol Biol Phys. 2001 Mar 15;49(4):917-30. doi: 10.1016/s0360-3016(00)01456-5. PMID 11240232
- [Background] Sonis ST, Elting LS, Keefe D, Peterson DE, Schubert M, Hauer-Jensen M, Bekele BN, Raber-Durlacher J, Donnelly JP, Rubenstein EB; Mucositis Study Section of the Multinational Association for Supportive Care in Cancer; International Society for Oral Oncology. Perspectives on cancer therapy-induced mucosal injury: pathogenesis, measurement, epidemiology, and consequences for patients. Cancer. 2004 May 1;100(9 Suppl):1995-2025. doi: 10.1002/cncr.20162. PMID 15108222
- [Background] Stokman MA, Spijkervet FK, Boezen HM, Schouten JP, Roodenburg JL, de Vries EG. Preventive intervention possibilities in radiotherapy- and chemotherapy-induced oral mucositis: results of meta-analyses. J Dent Res. 2006 Aug;85(8):690-700. doi: 10.1177/154405910608500802. PMID 16861284
- [Background] Worthington HV, Clarkson JE, Eden OB. Interventions for preventing oral mucositis for patients with cancer receiving treatment. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD000978. doi: 10.1002/14651858.CD000978.pub3. PMID 17943748
- [Background] Rothwell BR, Spektor WS. Palliation of radiation-related mucositis. Spec Care Dentist. 1990 Jan-Feb;10(1):21-5. doi: 10.1111/j.1754-4505.1990.tb01082.x. PMID 1689512
- [Background] Etiz D, Erkal HS, Serin M, Kucuk B, Hepari A, Elhan AH, Tulunay O, Cakmak A. Clinical and histopathological evaluation of sucralfate in prevention of oral mucositis induced by radiation therapy in patients with head and neck malignancies. Oral Oncol. 2000 Jan;36(1):116-20. doi: 10.1016/s1368-8375(99)00075-5. PMID 10889930
- [Background] Cengiz M, Ozyar E, Ozturk D, Akyol F, Atahan IL, Hayran M. Sucralfate in the prevention of radiation-induced oral mucositis. J Clin Gastroenterol. 1999 Jan;28(1):40-3. doi: 10.1097/00004836-199901000-00009. PMID 9916664